CLINICAL TRIAL: NCT03547713
Title: A Neuropsychological Characterization of Social Feedback Processing in Social Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: TASMC-18-TH-0082-17-TLV-CTIL
Record Dates: First submitted 2018-05-14; First posted 2018-06-06 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2018-05

CONDITIONS: Social Anxiety

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study group (Experimental): social feedback and neuropsychological assessment
  Interventions: Behavioral: Social feedback; Behavioral: Self-referential paradigm; Behavioral: Reward vs. punishment task; Behavioral: Emotional reactivity task

INTERVENTIONS:
Behavioral: Social feedback — Social feedback regarding performance of a public speech is delivered to participants
Behavioral: Self-referential paradigm — Exposure to traits varying in valence (positive vs. negative) and social domain (power vs. affiliation)
Behavioral: Reward vs. punishment task — Reception of monetary gains vs. losses
Behavioral: Emotional reactivity task — Exposure to emotional faces vs. shapes

SUMMARY:
The purpose of this study is to characterize neuropsychological mechanisms (positive affect, negative affect and self-evaluation) mediating processing of social feedback in people with different levels of social anxiety, by implementing functional and structural MRI.

DETAILED DESCRIPTION:
Social anxiety (SA) disorder is a relatively widespread emotional disorder which is associated with considerable impairment in social, educational, and occupational functioning (Kessler et al., 2005). This condition is characterized by a debilitating preoccupation with the evaluation of the self by others, ultimately leading to excessive fear and avoidance of interpersonal encounters. As opposed to healthy individuals who typically process social feedback in a positively biased manner, Individuals with high levels of SA tend to evaluate the feedback conveyed by others negatively. Such biases have a profound contribution to the maintenance of social-related concerns (Clark & Wells, 1995).

Thus, the overreaching goal of this research is to provide a neuropsychological account of biased processing of social feedback evident in SA. To meet this goal, participants varying in their level of SA are asked to deliver a speech and evaluate it before and after receiving social feedback during an fMRI scan. Additional structural and resting-state fMRI scans, as well as physiological and psychological measures, are obtained throughout the experiment in order to explain individual differences in processing of feedback. fMRI tasks probing basic neuropsychological processes include a self-referential paradigm, wherein participants judge if different traits varying in valence and social domain (power vs. affiliation) are descriptive of them; a reward vs. punishment task, in which participants can win or lose money; and an emotional reactivity task, in which participants view faces with different emotional expressions.

The long-term goal of this study is to better delineate both neurobiological and psychological models of SA, as well as to help in directing future neuromodulation-based treatments of mood and anxiety disorders.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants
* With different levels of social anxiety as measured by the Liebowitz Social Anxiety Scale-Self-Report (LSAS-SR; Fresco et al., 2001)
* Normal or corrected-to-normal vision
* Compatibility with general MRI requirements

Exclusion Criteria:

- History of neurological or psychiatric diseases

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2018-03-02 (Actual); Primary Completion 2018-10-23 (Actual); Study Completion 2018-10-23 (Actual)

PRIMARY OUTCOMES:
Change in evaluation of a public performance | 1 day
  Rating of a public performance made on a 0-10 scale before vs. after reception of social feedback
Correlation of social feedback processing with neural indices and anxiety levels | 1 day
  1. Neural activation and functional connectivity measured during processing of social feedback with different values.
  2. Neural activation and functional connectivity measured in fMRI tasks probing elemental neuropsychological processes:
  2.A. Processing of self-descriptive traits differing in valence (positive vs. negative) and social domain (power vs. affiliation).
  2.B. Response to emotional faces. 2.C. Anticipating and receiving monetary reward vs. loss. 3. Brain functional connectivity obtained during resting-state scans obtained at three time-points: a) before the speech; b) before feedback reception; c) after feedback reception.
  4. We will assess the correlation between multiple measurements (i.e. anxiety levels, behavioral indices of speech evaluation bias, and the battery of fMRI tasks) by implementing multivariate and multiparametric statistical models.

SECONDARY OUTCOMES:
Correlation of self-representation processes with neural indices and anxiety levels | 1 day
  1. Neural activation and functional connectivity measured during processing of social feedback with different values.
  2. Neural activation and functional connectivity measured in fMRI tasks probing elemental neuropsychological processes:
     b1. Processing of self-descriptive traits differing in valence (positive vs. negative) and social domain (power vs. affiliation).
     b2. Response to emotional faces. b3. Anticipating and receiving monetary reward vs. loss.
  3. Brain functional connectivity obtained during resting-state scans obtained at three time-points: before the speech, before feedback reception and after feedback reception.
  4. We will assess the correlation between multiple measurements (i.e. anxiety levels, behavioral indices of speech evaluation bias, and the battery of fMRI tasks) by implementing multivariate and multiparametric statistical models.

CONTACTS AND LOCATIONS:
Overall Officials: Talma Hendler, MD, Phd, Principal Investigator — Tel-Aviv Sourasky Medical Center
Locations (1):
- Tel-Aviv Sourasky medical center, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Fresco DM, Coles ME, Heimberg RG, Liebowitz MR, Hami S, Stein MB, Goetz D. The Liebowitz Social Anxiety Scale: a comparison of the psychometric properties of self-report and clinician-administered formats. Psychol Med. 2001 Aug;31(6):1025-35. doi: 10.1017/s0033291701004056. PMID 11513370
- [Background] Kessler RC, Chiu WT, Demler O, Merikangas KR, Walters EE. Prevalence, severity, and comorbidity of 12-month DSM-IV disorders in the National Comorbidity Survey Replication. Arch Gen Psychiatry. 2005 Jun;62(6):617-27. doi: 10.1001/archpsyc.62.6.617. PMID 15939839
- [Background] Clark, D. M., & Wells, A. (1995). A cognitive model of social phobia. Social Phobia: Diagnosis, Assessment, and Treatment, 41(68), 00022-3.